CLINICAL TRIAL: NCT04785352
Title: Grandi Byen: Supporting Child Growth and Development Through Integrated, Responsive Parenting, Nutrition and Hygiene
Brief Title: Grandi Byen: Test of an Integrated Parenting and Nutrition Intervention
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: Hôpital Universitaire Justinien (Unknown); Université Publique du Nord au Cap-Haïtien (Unknown); Konbit Sante (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Prevention
Other Study IDs: R01HD098255 (NIH)
Record Dates: First submitted 2021-02-24; First posted 2021-03-05 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Malnutrition, Child; Development, Child; Parenting
Keywords: Stunting; Responsive Parenting; Child Development
MeSH Terms: conditions — Child Nutrition Disorders; Growth Disorders | interventions — Diet Therapy

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: Raters assessing responsive parenting and child development outcomes will be blind to the condition of mother-child dyads.
  For investigators, they will be blinded to participants' assigned study arms before and during handling and analysis of the data.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Standard well-baby care (No Intervention): Children in this arm (control group), as well as children in the two intervention groups, will receive standard care as outlined in the Essential Package of Health Services by Haiti's Ministry of Public Health and Population (MSPP). This includes a World Health Organization (WHO) immunization schedule of vaccines, high dose vitamin A supplements, and growth monitoring and promotion.
- Nutrition Intervention (Experimental): Children in this arm will receive one egg per day for six months.
  Interventions: Dietary Supplement: Nutrition Intervention
- Grandi Byen (Experimental): This arm comprises a multicomponent intervention on responsive parenting, nutrition, hygiene, and one egg per day for six months for children.
  Interventions: Behavioral: Grandi Byen

INTERVENTIONS:
Dietary Supplement: Nutrition Intervention — One egg per day for six months
  Arms: Nutrition Intervention
Behavioral: Grandi Byen — Multicomponent intervention on responsive parenting, nutrition, hygiene + one egg per day for 6 months
  Arms: Grandi Byen

SUMMARY:
The premise of this trial is that a combined nutrition (eggs) and parenting behavior intervention (responsive parenting combined with the reinforcement of animal source foods and improved WASH) will synergistically result in improved child growth, development, and reduced enteric disease outcomes over and above a nutrition only intervention and standard well baby care.

This study is a 3-arm longitudinal randomized controlled trial (RCT) to compare the following groups for effectiveness in reducing young child stunted growth and enhancing overall development:1) standard well-baby care, (n=200); 2) nutrition intervention (one egg per day for 6 months), (n=200); and 3) multicomponent Grandi Byen intervention (responsive parenting, nutrition, hygiene + one egg per day for 6 months), (n=200).

Infants will be enrolled between 6-8 months of age and followed longitudinally for one year.

DETAILED DESCRIPTION:
A disturbingly high number of young children around the world experience stunted growth and development with irreparable consequences through the lifespan. Determinants of stunted growth and development are multi-factorial, including interactions between biological, behavioral, social, and environmental conditions, yet the evidence-base is minimal for integrated approaches to tackle the interwoven factors. Our group recently found significant impacts from an egg intervention on young child growth and biomarkers of nutrition and brain development. The effects on important psychosocial indicators of child development, however, were not assessed. Building on these findings and those of our pilot study of a group-based, multicomponent intervention (Grandi Byen, Haitian Creole for "grow well"), this randomized controlled trial (RCT) seeks to examine a greater breadth of egg intervention outcomes, the synergistic effects of adding psychoeducational parenting to the egg intervention, and mediating biological, behavioral and social factors.

The 3-arm longitudinal RCT will be carried out in Cap-Haitien, Haiti, where our group has a decade of research experience, established partnerships, and a strong research infrastructure. It is representative of resource-poor urban contexts globally, where parents face common economic and environmental challenges to child growth and development. The trial will compare the following groups for effectiveness in reducing young child stunted growth and enhancing overall development: 1) standard well-baby care, (n=200); 2) nutrition intervention (one egg per day for 6 months), (n=200); and 3) multicomponent Grandi Byen intervention (responsive parenting, nutrition, hygiene + one egg per day for 6 months), (n=200). Infants will be enrolled between 6-8 months of age and followed longitudinally for one year.

The specific aims of this project are:

Aim 1 (primary): To demonstrate the reproducibility and feasibility of egg-based interventions in reducing childhood stunting, and test its impact on development. Hypothesis 1: Linear growth will be increased by 0.30 LAZ in children receiving one egg per day compared to standard care. Hypothesis 2: Children receiving the egg intervention will have better cognitive, motor and language development compared to standard care. Question 1 (exploratory): Does an egg-based intervention impact social-emotional development?

Aim 2 (primary): To investigate the incremental benefit of Grandi Byen compared to egg only and standard care groups on primary outcomes of child growth and development. Hypothesis 3: Children of mothers receiving Grandi Byen will increase linear growth by 0.10 LAZ compared to the egg intervention. Hypothesis 4: Children of mothers receiving Grandi Byen will have higher scores on child cognition, language, motor, and socio-emotional development, with an effect size of 0.36 on cognition, compared to standard care. An economic evaluation will be conducted to compare the efficiency of the interventions.

Aim 3 (secondary). To explore pathways of intervention impacts on child growth and development by delineating the additive and synergistic effects of biological (nutrient biomarkers, bone age, and enteric disease), psychosocial (responsive parenting, cognitive stimulation), and environmental (hygiene and sanitation, diet) factors.

This study expands upon this earlier work by bringing together a transdisciplinary team spanning the biological and social sciences to work in partnership with Haitian collaborators. We will merge methods and concepts to produce comprehensive perspectives on several high priority areas including social, economic and biological factors that impact child brain development and function, nutrition among infants and very young children, determinants of bone health; and traumatic stress associated with growing up in abject poverty.

ELIGIBILITY:
Inclusion Criteria:

* Mothers/Caregivers 18 years or older of infants ages 6-8 months
* Infants ages 6-8 months
* Living in Petite Anse, Fort Saint Michel, Madeline, or similiar communities (Cap-Haitien, Haiti)

Exclusion Criteria:

* Multi-birth infant (twin, triplet, etc.)
* congenital health condition
* severe disabilities
* severely malnourished (WLZ<-3)
* child has an allergy to animal-source foods (specifically eggs, milk, or fish).

Ages: 6 Months to 8 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 600 (Actual)
Dates: Start 2021-07-01 (Actual); Primary Completion 2025-07-31 (Estimated); Study Completion 2025-07-31 (Estimated)

PRIMARY OUTCOMES:
Child Growth: Changes in length-for-age Z-score (LAZ) | Baseline and months 3, 6, 9, and 12
  Child length or height will be measured in centimeters (cm). Length-for-age Z-scores will be calculated using the World Health Organization (WHO) growth standards, accounting for the child sex and age in months.
Child Growth: Changes in weight-for-age Z-score (WAZ) | Baseline and months 3, 6, 9, and 12
  Child weight will be measured in kilograms (kg). Weight-for-age Z-scores will be calculated using the World Health Organization (WHO) growth standards, accounting for the child sex and age in months.
Child Growth: Changes in head circumference-for-age Z-score (HCZ) | Baseline and months 3, 6, 9, and 12
  Child head circumference will be measured in centimeters (cm). Head circumference-for-age Z-scores will be calculated using the World Health Organization (WHO) growth standards, accounting for the child sex and age in months.
Child Development: Changes in ASQ- Socio-Emotional (ASQ-SE) score | Baseline and months 6 and 12
  The Ages & Stages Questionnaire: Socio-Emotional Questionnaire (ASQ-SE2) will be used to assess and score child socio-emotional development.
Child Development: Changes in ASQ Communication score | Baseline and months 6 and 12
  The Ages & Stages Questionnaire (ASQ-3) will be used to assess and score children's communication skills.
Child Development: Changes in ASQ Gross Motor score | Baseline and months 6 and 12
  The Ages & Stages Questionnaire (ASQ-3) will be used to assess and score children's gross motor development.
Child Development: Changes in ASQ Fine Motor score | Baseline and months 6 and 12
  The Ages & Stages Questionnaire (ASQ-3) will be used to assess and score children's fine motor development.
Child Development: Changes in ASQ Problem Solving score | Baseline and months 6 and 12
  The Ages & Stages Questionnaire (ASQ-3) will be used to assess and score children's problem solving skills.

SECONDARY OUTCOMES:
Child Nutrient Biomarkers: Changes in Plasma Concentration of Docosahexaenoic acid (DHA) | Baseline and month 6
  Plasma concentration of DHA measured in µg/mL
Child Nutrient Biomarkers: Changes in Plasma Concentration of Choline | Baseline and month 6
  Plasma concentration of Choline measured in µg/mL
Child Nutrient Biomarkers: Changes in Plasma Concentration of Iron (Fe) | Baseline and month 6
  Plasma concentration of Iron (Fe) measured in mg/mL
Child Nutrient Biomarkers: Changes in Plasma Concentration of Zinc (Zn) | Baseline and month 6
  Plasma concentration of Zinc (Zn) measured in mg/mL
Child Nutrient Biomarkers: Changes in Plasma Concentration of Iodine (I) | Baseline and month 6
  Plasma concentration of Iodine (I) measured in mg/mL
Child Nutrient Biomarkers: Changes in Plasma Concentration of Selenium (Se) | Baseline and month 6
  Plasma concentration of Selenium (Se) measured in µg/mL
Child Bone Health: Changes in Bone Age Z-score | Baseline and months 3, 6, and 12
  Bone age z-scores are used as a measure of the child's bone health.
Child Dietary Intake | Baseline and months 6 and 12
  24-hour recalls and food frequency recalls are used to assess nutrient intakes, dietary diversity, and consumption of Animal-Source Foods (ASFs).
Responsive Parenting: Changes in PICCOLO Affection Score | Baseline and months 6 and 12
  Parenting Interactions with Children: Checklist of Observations Linked to Outcomes (PICCOLO) will be used to assess parent-child interactions, and a score for Affection will be calculated based on questionnaire items.
Responsive Parenting: Changes in PICCOLO Responsiveness Score | Baseline and months 6 and 12
  Parenting Interactions with Children: Checklist of Observations Linked to Outcomes (PICCOLO) will be used to assess parent-child interactions, and a score for Responsiveness will be calculated based on questionnaire items.
Responsive Parenting: Changes in PICCOLO Encouragement Score | Baseline and months 6 and 12
  Parenting Interactions with Children: Checklist of Observations Linked to Outcomes (PICCOLO) will be used to assess parent-child interactions, and a score for Encouragement will be calculated based on questionnaire items.
Responsive Parenting: Changes in HOME Scores | Baseline and months 6 and 12
  The Home Observation Measurement of the Environment (HOME) inventory will be used in assessing the home environment.
Child Morbidities | Baseline and months 3, 6, 9, 12
  Diarrhea, respiratory conditions, allergies.

CONTACTS AND LOCATIONS:
Overall Officials: Lora L Iannotti, PhD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Hôpital Universitaire Justinien, Cap-Haïtien, Haiti

IPD SHARING:
Plan to Share IPD: Yes
Data collected for this study will be analyzed and stored on the on the REDCap platform and on Box, a secure, HIPAA and FERPA compliant data storage and online sharing platform. After the study is completed, the de-identified, archived data will be transmitted to and stored in a secure folder on Box; other researchers, including those outside of the study, who would want to use the deidentified data will only be able to access the data following approval from the PIs. Information pertaining to data sharing with other researchers is detailed during the informed consent process.
  During the conduct of the study, an individual participant can choose to withdraw consent to have biological specimens stored for future research. However, withdrawal of consent with regard to biosample storage may not be possible after the study is completed.
  When the study is completed, access to study data and/or samples will be provided through the approval of the PIs.
Supporting Information: Study Protocol, SAP, ICF
Access Criteria: Researchers wanting to use the data would have to contact the PIs and explain their purpose for using the data.

REFERENCES:
- [Derived] Kohl PL, Gyimah EA, Diaz J, Kuhlmann FM, Dulience SJ, Embaye F, Brown DS, Guo S, Luby JL, Nicholas JL, Turner J, Chapnick M, Pierre JM, Boncy J, St Fleur R, Black MM, Iannotti LL. Grandi Byen-supporting child growth and development through integrated, responsive parenting, nutrition and hygiene: study protocol for a randomized controlled trial. BMC Pediatr. 2022 Jan 21;22(1):54. doi: 10.1186/s12887-021-03089-x. PMID 35062907